CLINICAL TRIAL: NCT01311089
Title: A Comparative Study of Robotic Thyroidectomy Using Transaxillary Approach Versus Conventional Open Thyroidectomy : Postoperative Body Image Change and Cosmetic Satisfaction
Brief Title: A Comparative Study of Robotic Thyroidectomy Using Transaxillary Approach Versus Conventional Open Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2010-0055
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Papillary Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic thyroidectomy group: Robotic thyroidectomy group is the patient group who underwent robot-assisted endoscopic thyroid surgery using a gasless, trans-axillary approach.
- conventional open thyroidectomy group: Conventional open thyroidectomy group is th patient group who underwent thyroid surgery via neck incision.

SUMMARY:
Most patients with thyroid tumors are effectively treated surgically by practitioners experienced in the techniques of thyroidectomy. Many patients, especially women, undergoing thyroid surgery are concerned about the postoperative cosmetic appearance of the neck. Robotic thyroidectomy which can hide the operative scar was associated with a higher degree of patient cosmetic satisfaction.

DETAILED DESCRIPTION:
Most patients with thyroid tumors are effectively treated surgically by practitioners experienced in the techniques of thyroidectomy. Many patients, especially women, undergoing thyroid surgery are concerned about the postoperative cosmetic appearance of the neck. Robotic thyroidectomy which can hide the operative scar was associated with a higher degree of patient cosmetic satisfaction. In this study, we designed a prospective study comparing the cosmetic satisfaction and the postoperative body image change which associated with patient self-esteem between robotic thyroidectomy and conventional open thyroidectomy group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with papillary thyroid carcinoma who underwent thyroidectomy
* Age was over 20 years old

Exclusion Criteria:

* Keloid
* Previous neck or anterior chest operation history
* The patients who underwent combined radical neck dissection
* The patient with postoperative wound problem
* The patient with underlying systemic disease which can make influences on the wound healing process
* The patient who can not read and understand the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients with papillary thyroid carcinoma who underwent thyroidectomy at Yonsei University Health System were enrolled. 60patients were conventional open thyroidectomy group and 60 patients were robotic thyroidectomy group. All of these patients was over 20 years old.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Tan CT, Cheah WK, Delbridge L. "Scarless" (in the neck) endoscopic thyroidectomy (SET): an evidence-based review of published techniques. World J Surg. 2008 Jul;32(7):1349-57. doi: 10.1007/s00268-008-9555-3. PMID 18360737
- [Background] Kang SW, Lee SC, Lee SH, Lee KY, Jeong JJ, Lee YS, Nam KH, Chang HS, Chung WY, Park CS. Robotic thyroid surgery using a gasless, transaxillary approach and the da Vinci S system: the operative outcomes of 338 consecutive patients. Surgery. 2009 Dec;146(6):1048-55. doi: 10.1016/j.surg.2009.09.007. Epub 2009 Oct 30. PMID 19879615
- [Background] Jeong JJ, Kang SW, Yun JS, Sung TY, Lee SC, Lee YS, Nam KH, Chang HS, Chung WY, Park CS. Comparative study of endoscopic thyroidectomy versus conventional open thyroidectomy in papillary thyroid microcarcinoma (PTMC) patients. J Surg Oncol. 2009 Nov 1;100(6):477-80. doi: 10.1002/jso.21367. PMID 19653245
- [Background] Kang SW, Jeong JJ, Nam KH, Chang HS, Chung WY, Park CS. Robot-assisted endoscopic thyroidectomy for thyroid malignancies using a gasless transaxillary approach. J Am Coll Surg. 2009 Aug;209(2):e1-7. doi: 10.1016/j.jamcollsurg.2009.05.003. Epub 2009 Jun 12. No abstract available. PMID 19632588
- [Background] Chung YS, Choe JH, Kang KH, Kim SW, Chung KW, Park KS, Han W, Noh DY, Oh SK, Youn YK. Endoscopic thyroidectomy for thyroid malignancies: comparison with conventional open thyroidectomy. World J Surg. 2007 Dec;31(12):2302-6; discussion 2307-8. doi: 10.1007/s00268-007-9117-0. PMID 17566819
- [Background] Yoon JH, Park CH, Chung WY. Gasless endoscopic thyroidectomy via an axillary approach: experience of 30 cases. Surg Laparosc Endosc Percutan Tech. 2006 Aug;16(4):226-31. doi: 10.1097/00129689-200608000-00006. PMID 16921301
- [Background] Inukai M, Usui Y. Clinical evaluation of gasless endoscopic thyroid surgery. Surg Today. 2005;35(3):199-204. doi: 10.1007/s00595-004-2929-8. PMID 15772789
- [Background] Ohgami M, Ishii S, Arisawa Y, Ohmori T, Noga K, Furukawa T, Kitajima M. Scarless endoscopic thyroidectomy: breast approach for better cosmesis. Surg Laparosc Endosc Percutan Tech. 2000 Feb;10(1):1-4. PMID 10872517
- [Background] Ikeda Y, Takami H, Sasaki Y, Takayama J, Niimi M, Kan S. Comparative study of thyroidectomies. Endoscopic surgery versus conventional open surgery. Surg Endosc. 2002 Dec;16(12):1741-5. doi: 10.1007/s00464-002-8830-x. Epub 2002 Jul 29. PMID 12140635
- [Background] Lee J, Nah KY, Kim RM, Ahn YH, Soh EY, Chung WY. Differences in postoperative outcomes, function, and cosmesis: open versus robotic thyroidectomy. Surg Endosc. 2010 Dec;24(12):3186-94. doi: 10.1007/s00464-010-1113-z. Epub 2010 May 19. PMID 20490558